CLINICAL TRIAL: NCT01350245
Title: A Two Step Approach to Allogeneic Hematopoietic Stem Cell Transplantation for Patients With Hematologic Malignancies in Remission From HLA Partially-Matched Related Donors
Brief Title: Bone Marrow Transplantation of Patients in Remission Using Partially Matched Relative Donor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10D.219; 2010-10 (Other: CCRRC); JT 2150 (Other: JeffTrial Number)
Record Dates: First submitted 2011-05-04; First posted 2011-05-09 (Estimated); Results first posted 2014-10-13 (Estimated); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes; Biphenotypic Leukemia; Acute Lymphocytic Leukemia; Chronic Myeloid Leukemia; Chronic Lymphocytic Leukemia; Plasma Cell Neoplasms; Lymphoma; Hodgkin's Disease; Aplastic Anemia
Keywords: Acute Myeloid Leukemia; Myelodysplastic Syndromes; Biphenotypic Leukemia; Acute Lymphocytic Leukemia; Chronic Myeloid Leukemia; Chronic Lymphocytic Leukemia; Plasma Cell Neoplasms; Lymphoma; Hodgkin's Disease; Aplastic Anemia; Hematopoietic stem cell transplant (HSCT); myeloablative haploidentical HSCT; graft versus host disease (GVHD)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Lymphocytic, Chronic, B-Cell; Neoplasms, Plasma Cell; Lymphoma; Hodgkin Disease; Anemia, Aplastic; Graft vs Host Disease | interventions — Whole-Body Irradiation; Cyclophosphamide; Mycophenolic Acid; Tacrolimus; Hematopoietic Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TJU 2 Step Regimen (Experimental): All patients treated on this trial will have hematological malignancies that are in remission at the time of the transplant. Their diseases would be expected to relapse with standard therapy alone.
  Interventions: Radiation: Total Body Irradiation (TBI); Biological: Donor Lymphocyte Infusion (DLI); Drug: Cyclophosphamide; Drug: Mycophenolate Mofetil (MMF); Drug: Tacrolimus; Device: Hematopoietic stem cell transplantation (HSCT)

INTERVENTIONS:
Radiation: Total Body Irradiation (TBI) — Total body irradiation is given in 8 fractions over 4 days (total dose of 12 Gy).
Biological: Donor Lymphocyte Infusion (DLI) — After TBI, the patients will receive a dose of 2 x 10e8 of their donor's T cells. After this infusion, the patients will have 2 rest days.
Drug: Cyclophosphamide — Cyclophosphamide is administered 2 days after the DLI to help tolerize the donor T cells. It is given at a dose of 60 mg/kg/d for 2 days
  Other Names: Endoxan; Cytoxan; Neosar; Procytox; Revimmune; cytophosphane
Drug: Mycophenolate Mofetil (MMF) — Started the day before the transplant to prevent graft versus host disease (GVHD)
  Other Names: CellCept
Drug: Tacrolimus — Started the day before the transplant to prevent graft-versus-host disease (GVHD)
  Other Names: FK-506; Fujimycin
Device: Hematopoietic stem cell transplantation (HSCT) — One day after the cyclophosphamide is finished, the patients will receive a CD34 selected-donor stem cell product. This is the day of transplant.
  The CliniMACS® Plus Instrument will be used for the selection of human CD34+ hematopoietic stem and progenitor cells in human allogeneic hematopoietic stem cell transplantation.
  Other Names: CliniMACS

SUMMARY:
The primary hypothesis of this research study is that patients in remission undergoing myeloablative haploidentical hematopoietic stem cell transplantation (HSCT) on the Thomas Jefferson University (TJU) 2 Step treatment regimen will have a disease-free survival (DFS) rate at 1 year that is the same or better than the historical DFS of patients with similar diagnoses and ages undergoing matched sibling HSCT. Based on a review of the literature a DFS rate of 50% or better at 1 year would meet the criterion for an effective alternative therapy. A DFS rate of 75% or better would imply superior efficacy of the TJU 2 Step approach over T-replete matched sibling HSCT.

DETAILED DESCRIPTION:
The primary rationale for the development of this research study is to find out if the Thomas Jefferson University (TJU) 2 Step approach to stem cell transplant is an effective treatment for patients with blood cancers who require transplant for long-term survival but are without an available matched-sibling donor. Historically, survival rates for patients undergoing half-matched stem cell transplant have been much lower than those observed after matched sibling stem cell transplant. This may be due to the poor-risk disease features of the patients by the time they are referred for hematopoietic stem cell transplantation (HSCT). Survival post half-matched stem cell transplant has also been affected by the requirement to remove or soothe donor T cells resulting in higher rates of infection and relapse. Newer approaches to haploidentical HSCT, such as the TJU 2 Step approach, utilize cyclophosphamide (CY) to tolerize donor lymphocytes instead of removing them completely from the donor product. This has resulted in less infection without concomitant increase in severe graft-versus-host disease (GVHD) and has increased overall survival as compared to older haploidentical treatment approaches due to decreases in regimen-related morbidity.

Because of the historically low overall survival (OS) after haploidentical HSCT, it has become a procedure of last resort with most centers unwilling to consider it unless all other options are exhausted. With the recent development of regimens such as the TJU 2 Step approach which provide safe, alternative platforms for HSCT, it is now feasible, and ethically more acceptable, for patients without matched sibling donors to undergo HSCT prior to being heavily pretreated or developing resistant disease. In this setting, i.e. equivalent regimen safety profiles and more homogenous patient comparison groups, it is possible to more accurately compare antitumor effects between matched sibling donors and haploidentical donors. There is ample evidence in the literature that HLA mismatching causes GVHD. There is not a large body of evidence supporting the notion that HLA mismatching provides superior tumor control translating into greater relapse free survival. As compared to more common types of transplants where donor T cells are given to the recipient, the investigators would surmise that the T cell tolerization associated with the TJU 2 Step approach may decrease the anti-tumor effects of the donor immune system. Conversely, the greater degree of human leukocyte antigen (HLA) mismatch with exploitation of NK effects may mitigate some of the attenuated T cell alloreactivity.

Thus, in the context of comparable regimen-related toxicity, our major aim in this research study is to compare graft versus tumor effects as measured by disease-free survival (DFS) between matched sibling HSCT and the TJU 2 Step haploidentical HSCT. If DFS is similar despite T cell tolerization, than the TJU 2 Step haploidentical approach should be considered an effective alternative therapy for those patients in remission without a matched sibling donor. The widespread benefit of this outcome would be the enfranchisement of segments of the population who are without available matched donors resulting in a delay or a failure to receive this potentially life-saving therapy. If DFS survival after treatment on the TJU 2 Step haploidentical approach is superior to what would be expected after matched sibling HSCT, then one could conclude that haploidentical HSCT confers greater tumor control forming the basis for future studies regarding the potential benefits of utilizing haploidentical donors over matched sibling donors when both types of donors are available.

ELIGIBILITY:
Inclusion Criteria:

1. Any patient with a hematologic or oncologic diagnosis without morphological evidence of disease in which allogeneic HSCT is thought to be beneficial.

   * Diagnoses include:

   Acute Myeloid Leukemia Myelodysplastic Syndromes Biphenotypic Leukemia Acute Lymphocytic Leukemia Chronic Myeloid Leukemia Chronic Lymphocytic Leukemia Plasma Cell Neoplasms Lymphoma Hodgkin Disease Aplastic Anemia
2. Patients must have a related donor who is a two or more allele mismatch at the HLA-A; B; C; DR loci.
3. Patients must adequate organ function:

   * LVEF of > or = 50%
   * DLCO > or = 50% of predicted corrected for hemoglobin
   * Adequate liver function as defined by a serum bilirubin < or = 1.8, AST or ALT < or = 2.5X upper limit of normal
   * Creatinine clearance of > or = 60 ml/min
4. Performance status > or = 70% (TJU Karnofsky)
5. HCT-CI Score < 5 Points
6. Patients must be willing to use contraception if they have childbearing potential
7. Able to give informed consent

Exclusion Criteria:

1. Performance status < or = 70% (TJU Karnofsky)
2. HCT-CI Score > 5 Points
3. Combination of Performance status of < 80% (TJU Karnofsky) and an HCT-CI of 4 points or more.
4. HIV positive
5. Active involvement of the central nervous system with malignancy
6. Psychiatric disorder that would preclude patients from signing an informed consent
7. Pregnancy
8. Patients with life expectancy of < or = 6 months for reasons other than their underlying hematologic/oncologic disorder
9. Patients who have received alemtuzumab within 8 weeks of the transplant admission, or who have recently received horse or rabbit ant-thymocyte globulin and have an ATG level of > or = 2 ugm/ml
10. Patients who cannot receive cyclophosphamide
11. Patients with evidence of another malignancy, exclusive of a skin cancer that requires only local treatment, should not be enrolled on this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-07; Primary Completion 2013-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dolores Grosso, DNP, CRNP, Principal Investigator — Thomas Jefferson University; Neal Flomenberg, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Kimmel Cancer Center at Thomas Jefferson University, an NCI-Designated Cancer Center — http://www.KimmelCancerCenter.org
- See also: Thomas Jefferson University Hospitals — http://www.JeffersonHospital.org

RESULTS

PARTICIPANT FLOW:
Groups:
- TJU 2 Step Regimen: All patients treated on this trial will have hematological malignancies that are in remission at the time of the transplant. Their diseases would be expected to relapse with standard therapy alone.
  Total Body Irradiation (TBI): Total body irradiation given in 8 fractions over 4 days (total dose of 12 Gy).
  Donor Lymphocyte Infusion (DLI): After TBI, the patients will receive a dose of 2 x 10e8 of their donor's T cells. After this infusion, the patients will have 2 rest days.
  Cyclophosphamide: Cyclophosphamide is administered 2 days after the DLI to help tolerize the donor T cells. It is given at a dose of 60 mg/kg/d for 2 days
  Mycophenolate Mofetil (MMF): Started the day before the transplant to prevent graft versus host disease (GVHD)
  Tacrolimus: Started the day before the transplant to prevent graft-versus-host disease (GVHD)
  Hematopoietic stem cell transplantation (HSCT): One day after the cyclophosphamide is finished, the patients will receive a CD34 selected-do
Period: Overall Study
Arm/Group | TJU 2 Step Regimen
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | TJU 2 Step Regimen
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.2 (14.3)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 22
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Disease-Free Survival (DFS)
Description: 1-year post-transplant disease free survival (DFS), defined as success if a patient is alive and disease free at 1-year post-transplant.
Time Frame: 1 year post-transplant
Measure: Number; unit: percentage of patients
Arm/Group | TJU 2 Step Regimen
Number analyzed (Participants) | 28
percentage of patients | 78.6

2. Primary Outcome: Probability of Overall Survival at 15 Months Post-treatment
Description: Probability of overall survival at 15 months post-treatment, defined as success if a patient is alive 1-year post-transplant.
Time Frame: 15 months
Measure: Number; unit: percentage of probability
Arm/Group | TJU 2 Step Regimen
Number analyzed (Participants) | 28
percentage of probability | 85

ADVERSE EVENTS:
Arm/Group | TJU 2 Step Regimen
Serious Adverse Events (participants affected / at risk) | 19/28
Other Adverse Events (participants affected / at risk) | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TJU 2 Step Regimen (N=28)
Bone marrow cellularity (Musculoskeletal and connective tissue disorders) | 1 (1)
Infection (General disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Fever (General disorders) | 8 (10)
Headache (General disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
CMV reactivation (Immune system disorders) | 4 (4)
BK cystitis (General disorders) | 1 (1)
Nausea (General disorders) | 1 (1)
HHV-6 infection (Blood and lymphatic system disorders) | 2 (2)
Subdural hematoma (Skin and subcutaneous tissue disorders) | 1 (1)
Brain injury from subdural hematoma (Skin and subcutaneous tissue disorders) | 1 (1)
Sepsis (Blood and lymphatic system disorders) | 1 (1)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cholecystitis (Gastrointestinal disorders) | 1 (1)
Hypoxia (General disorders) | 2 (2)
Acute infusion reaction (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TJU 2 Step Regimen (N=28)
Headache (General disorders) | 18 (30)
Decreased appetite (General disorders) | 7 (7)
Anxiety (Psychiatric disorders) | 19 (22)
Rigors (General disorders) | 7 (8)
Tachycardia (Cardiac disorders) | 20 (35)
Malaise (General disorders) | 2 (2)
Oral discomfort (General disorders) | 1 (1)
Sore throat (General disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 23 (52)
Ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 26 (27)
Back pain (General disorders) | 13 (16)
Insomnia (General disorders) | 18 (21)
Dry mouth (General disorders) | 11 (12)
Hallucinations (Psychiatric disorders) | 2 (2)
Parasthesia of foot (Nervous system disorders) | 2 (2)
Dysphagia (General disorders) | 3 (3)
Tongue sores (Skin and subcutaneous tissue disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Epigastric pain/heartburn (Gastrointestinal disorders) | 9 (11)
Odynophagia (General disorders) | 1 (1)
Alopecia (General disorders) | 1 (1)
Clubbing of extremities (General disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2)
Gum pain at site of tooth extraction (General disorders) | 1 (1)
Itching (General disorders) | 10 (12)
Hypertension (Blood and lymphatic system disorders) | 12 (16)
Cheek pain (General disorders) | 1 (1)
Jaw pain (General disorders) | 3 (3)
Nausea (General disorders) | 11 (13)
Leg pain (General disorders) | 6 (6)
Swollen eyelid (General disorders) | 1 (1)
Hand pain (General disorders) | 2 (2)
Abdominal pain (General disorders) | 17 (25)
Numbness/tingling (Nervous system disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 25 (58)
Constipation (Gastrointestinal disorders) | 13 (19)
Congestion (Respiratory, thoracic and mediastinal disorders) | 11 (14)
Cold-like symptoms (General disorders) | 2 (2)
Flushing/erythema (Skin and subcutaneous tissue disorders) | 2 (2)
Mucositis (Gastrointestinal disorders) | 24 (24)
Hyperbilirubinemia (Blood and lymphatic system disorders) | 7 (9)
Vision - flashing lights (Eye disorders) | 1 (1)
Vomiting (General disorders) | 2 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 10 (12)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
Mild desquamation on fingers (Skin and subcutaneous tissue disorders) | 1 (1)
Knee - decreased range of motion (Musculoskeletal and connective tissue disorders) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Plaque on tongue (General disorders) | 1 (1)
Fever (General disorders) | 24 (58)
Hypotension (Blood and lymphatic system disorders) | 19 (28)
Vasovagal syncope (General disorders) | 2 (2)
Dizziness/lightheaded (General disorders) | 12 (16)
Dysuria (Renal and urinary disorders) | 10 (13)
Tremors (General disorders) | 6 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 15 (23)
General pain (General disorders) | 3 (3)
Pain at PICC site (General disorders) | 2 (2)
Anorexia (General disorders) | 8 (8)
Sweats (General disorders) | 3 (3)
Blurry vision (Eye disorders) | 4 (4)
Night sweats (General disorders) | 1 (1)
Chills (General disorders) | 8 (11)
Abdominal cramps (General disorders) | 3 (3)
Cytomegalovirus reactivation (General disorders) | 5 (5)
Hip pain (General disorders) | 4 (4)
Decreased sense of well-being (Psychiatric disorders) | 1 (1)
Hypokalemia (Blood and lymphatic system disorders) | 3 (4)
Muscle pain (General disorders) | 8 (8)
Puffy face (General disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 7 (7)
Hyponatremia (General disorders) | 5 (6)
Leg cramping (General disorders) | 1 (1)
Perinephric fluid (Renal and urinary disorders) | 1 (1)
Head cold (General disorders) | 1 (1)
Clostridium difficile (Gastrointestinal disorders) | 6 (8)
Depression (Psychiatric disorders) | 7 (7)
Nocturia (Renal and urinary disorders) | 9 (9)
Muscle weakness (General disorders) | 1 (1)
Hearing problems (Ear and labyrinth disorders) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Neuropathy (Nervous system disorders) | 7 (7)
Edema (Skin and subcutaneous tissue disorders) | 4 (4)
Diminished breath sounds (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Knee pain (General disorders) | 3 (3)
Decreased urine output (Renal and urinary disorders) | 7 (8)
BK viremia (Renal and urinary disorders) | 1 (1)
Visual acuity change/weakness (Eye disorders) | 3 (3)
Papules (Skin and subcutaneous tissue disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 3 (3)
Groin pain (General disorders) | 1 (1)
Heel/ankle pain (General disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Ventricular systolic dysfunction (Cardiac disorders) | 3 (3)
Hematuria (Renal and urinary disorders) | 2 (2)
Trouble sleeping (General disorders) | 7 (9)
Lethargic (General disorders) | 11 (11)
Hypoxia (General disorders) | 6 (9)
Dry eyes (Eye disorders) | 3 (3)
Dry cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Mouth ulceration (General disorders) | 1 (1)
Nose dryness (General disorders) | 1 (1)
Fluid overload (Blood and lymphatic system disorders) | 7 (8)
Increased creatinine (Blood and lymphatic system disorders) | 7 (10)
Hiccups (General disorders) | 3 (3)
Burning of soles of hands and feet (Skin and subcutaneous tissue disorders) | 1 (1)
Ear pain (General disorders) | 4 (4)
Shoulder pain (General disorders) | 4 (4)
Eye pain (General disorders) | 1 (1)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Bloated feeling (General disorders) | 2 (2)
Arm swelling (General disorders) | 4 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Retinal hemorrhage (Eye disorders) | 2 (2)
Increased LFTs (Hepatobiliary disorders) | 4 (6)
Neck pain (General disorders) | 2 (3)
Mild distress (Psychiatric disorders) | 1 (1)
Pericather thrombus (Blood and lymphatic system disorders) | 3 (3)
Frustration (Psychiatric disorders) | 1 (1)
Meningitis (Infections and infestations) | 1 (1)
Photophobia (Eye disorders) | 3 (3)
Urinary incontinence (Renal and urinary disorders) | 3 (3)
Orange urine (Renal and urinary disorders) | 1 (1)
Seizures (Nervous system disorders) | 1 (2)
Pericardial effusion (Cardiac disorders) | 6 (6)
Hypernatremia (Blood and lymphatic system disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Abdominal distension (Skin and subcutaneous tissue disorders) | 1 (1)
Penile lesion (Skin and subcutaneous tissue disorders) | 1 (2)
Bradycardia (Cardiac disorders) | 2 (3)
Polyuria (Renal and urinary disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Agitation (Psychiatric disorders) | 2 (3)
Internal jugular thrombus (Blood and lymphatic system disorders) | 1 (1)
Opisthotonus (Musculoskeletal and connective tissue disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Blisters (Skin and subcutaneous tissue disorders) | 1 (1)
Enlarged lymph node (General disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Gastroparesis pain (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 8 (10)
Indigestion (Gastrointestinal disorders) | 1 (1)
Neck stiffness (General disorders) | 3 (6)
Orthostatic hypotension (Blood and lymphatic system disorders) | 2 (2)
Neutropenic colitis (Gastrointestinal disorders) | 1 (1)
Ringing in ears (Ear and labyrinth disorders) | 1 (1)
Hyperglycemia (Blood and lymphatic system disorders) | 2 (2)
Altered mental status (Psychiatric disorders) | 2 (2)
Hypoglycemia (Blood and lymphatic system disorders) | 1 (1)
HHV-6 reactivation (Blood and lymphatic system disorders) | 2 (2)
Hypomagnesemia (Blood and lymphatic system disorders) | 1 (1)
Hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Speech or memory change (Psychiatric disorders) | 1 (1)
Sensitivity to hot/cold (Nervous system disorders) | 1 (1)
Swollen face (General disorders) | 1 (1)
Electrolyte imbalance (Blood and lymphatic system disorders) | 9 (9)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1)
Pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pain at lung biopsy site (General disorders) | 1 (1)
Difficulty walking (General disorders) | 1 (1)
Feet pain (General disorders) | 3 (3)
Malnutrition (General disorders) | 1 (1)
Weight loss (General disorders) | 1 (1)
Platelet infusion reaction (Blood and lymphatic system disorders) | 1 (1)
Hot flashes (General disorders) | 1 (1)
Auditory hallucinations (Psychiatric disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 3 (3)
Elevated ferritin (Blood and lymphatic system disorders) | 1 (1)
Arm pain (General disorders) | 3 (5)
Tearing of eyes (Eye disorders) | 1 (1)
Swollen ankles (General disorders) | 1 (1)
Thrush (Infections and infestations) | 2 (2)
Urinary retention (Renal and urinary disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dehydration (General disorders) | 2 (2)
Volume overload (Cardiac disorders) | 1 (1)
Hives (Skin and subcutaneous tissue disorders) | 2 (2)
Hypercholesterolemia (Blood and lymphatic system disorders) | 1 (1)
Vagina - whitish coating (Reproductive system and breast disorders) | 1 (1)
Hyperlipidemia (Blood and lymphatic system disorders) | 2 (2)
Bone pain (General disorders) | 2 (3)
Discouraged (Psychiatric disorders) | 1 (1)
Blindness (Eye disorders) | 1 (1)
Penile/scrotum pain (General disorders) | 1 (1)
Penile blister (Skin and subcutaneous tissue disorders) | 1 (1)
Tongue lumps (General disorders) | 1 (1)
Nightmares (Psychiatric disorders) | 1 (1)
Altered taste (General disorders) | 1 (1)
Parotitis (General disorders) | 1 (1)
Difficulty concentrating (General disorders) | 1 (1)
Visual disturbance (General disorders) | 1 (1)
Shin pain (General disorders) | 1 (1)
Joint aches (Musculoskeletal and connective tissue disorders) | 1 (1)
Low TSH (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes